CLINICAL TRIAL: NCT03234231
Title: Supervised Toothbrushing Programme and Oral Health Education for Intellectual Disabled Students: A Cluster Randomised Controlled Trial
Brief Title: Supervised Brushing Programme for Intellectual Disabled Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MD Equation (Industry)
Responsible Party: Principal Investigator, Cecilia Young, Founder, MD Equation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HM01
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Oral Health; Intellectual Disability; Randomized Controlled Trial
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: data entered by independent clerical staff with no information of the detail of the study outcomes assessor will not be told which group of subjects are examined but there is a chance that the subjects tell him/her
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group receive nothing during the study period.
- Intervention Group (Experimental): A 3-month supervised tooth brushing programme will be provided to the students. An oral health education talk with written material delivered to the carers and the students
  Interventions: Behavioral: 3-month supervised tooth brushing programme; Behavioral: oral health education talk

INTERVENTIONS:
Behavioral: 3-month supervised tooth brushing programme — One or a few dental hygienists, who are trained to teach how to brush and provide scaling, will supervise the students to brush daily in school for three months.
  Arms: Intervention Group
Behavioral: oral health education talk — It is conducted by a dentist, while written materials will be delivered to the students and their carers.
  Arms: Intervention Group

SUMMARY:
Intellectual disabled persons faced more dental problems. According to a medical review paper of international and local studies, this group has poorer dental hygiene, more severe gum disease and more untreated caries. In 2010, a report from the guardians in Hong Kong mentioned that most adults with intellectual disability cannot clean their teeth, the have dental problems and it is very difficult for intellectually disabled students to co-operate during the dental treatment. In order to alleviate their dental problems, supervised toothbrushing programme and an oral health education talk are proposed. The investigators investigate the effectiveness of the supervised toothbrushing programme and an oral health education talk. The target group of the study is mild to moderate grade intellectual disabled students of special schools in Hong Kong. A clustered randomised controlled trial design is adopted.

DETAILED DESCRIPTION:
Intellectual disabled persons faced more dental problems. According to a medical review paper of international and local studies, this group has poorer dental hygiene, more severe gum disease and more untreated caries. In 2010, a report from the guardians in Hong Kong mentioned that most adults with intellectual disability cannot clean their teeth, the have dental problems and it is very difficult for intellectually disabled students to co-operate during the dental treatment. In order to alleviate their dental problems, supervised toothbrushing programme and an oral health education talk are proposed. The investigators investigate the effectiveness of the supervised toothbrushing programme and an oral health education talk. The target group of the study is mild to moderate grade intellectual disabled students of special schools in Hong Kong. A clustered randomised controlled trial design is adopted.

ELIGIBILITY:
Inclusion Criteria:

* Mild and moderate grade intellectual disabled students in special schools.

Exclusion Criteria:

* 1. Those students who have simultaneously joined other oral health programme during the study period.
* 2. Those students with the presence of conditions rendering a need of antibiotic prophylaxis prior to periodontal examination e.g. rheumatic heart disease.
* 3. Uncooperative students that oral examination is not possible.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 602 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Gingivitis score | A study period of 3 months
  Measuring the change of oral conditions of the students

SECONDARY OUTCOMES:
Plaque score | A study period of 3 months
  Measuring the change of oral conditions of the students

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Young, BDS(HK),MPH, Principal Investigator — MD Equation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anders PL, Davis EL. Oral health of patients with intellectual disabilities: a systematic review. Spec Care Dentist. 2010 May-Jun;30(3):110-7. doi: 10.1111/j.1754-4505.2010.00136.x. PMID 20500706
- [Background] Stefanovska E, Nakova M, Radojkova-Nikolovska V, Ristoska S. Tooth-brushing intervention programme among children with mental handicap. Bratisl Lek Listy. 2010;111(5):299-302. PMID 20568423
- [Background] Shyama M, Al-Mutawa SA, Honkala S, Honkala E. Supervised toothbrushing and oral health education program in Kuwait for children and young adults with Down syndrome. Spec Care Dentist. 2003;23(3):94-9. doi: 10.1111/j.1754-4505.2003.tb01668.x. PMID 14650557
- [Background] Rabe-Jablonska J, Bienkiewicz W. [Anxiety disorders in the fourth edition of the classification of mental disorders prepared by the American Psychiatric Association: diagnostic and statistical manual of mental disorders (DMS-IV -- options book]. Psychiatr Pol. 1994 Mar-Apr;28(2):255-68. Polish. PMID 8208869
- See also: A report from the guardians in Hong Kong mentioned that most adults with intellectual disability cannot clean their teeth, the have dental problems and it is very difficult for them to co-operate during the dental treatment. (Chinese only) — http://www.hkjcpmh.org.hk/uploads/books/pdf/178344fa63dc4fa193b998268e345219.pdf